CLINICAL TRIAL: NCT00353405
Title: A Multilevel HIV Prevention Strategy for High-Risk Youth
Brief Title: HIV and STD Prevention for High-Risk, Inner-City, African American Youth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Daniel Romer, Director, Adolescent Risk Communication Institute, Annenberg Public Policy Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U01MH066809 (NIH); U01MH066809 (NIH); DAHBR 9A-ASAC
Record Dates: First submitted 2006-07-14; First posted 2006-07-18 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: Adolescents; Sexually Transmitted Infections; Gonorrhea; Chlamydia Infections
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Gonorrhea; Chlamydia Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants receiving social skills training and mass media messages
  Interventions: Behavioral: Social Skills Training; Behavioral: Mass media
- 2 (Experimental): Participants receiving social skills training and no mass media messages
  Interventions: Behavioral: Social Skills Training
- 3 (Experimental): Participants receiving mass media messages and no social skills training
  Interventions: Behavioral: Mass media
- 4 (Experimental): Participants receiving no social skills training and no mass media messages
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Social Skills Training — Social skills training includes two 8-hour sexual health skills building sessions conducted in the community.
  Arms: 1; 2
Behavioral: Mass media — Mass media provides messages that support sexual health skills.
  Arms: 1; 3
Behavioral: Control — Control group received no social skills training and no media mass media messages.
  Arms: 4

SUMMARY:
This study will evaluate the joint and separate effectiveness of two HIV/STD prevention programs in providing protection against acquiring STDs and maintaining safer sex behavior.

DETAILED DESCRIPTION:
Approximately 25% of the new HIV cases in the United States each year occur among adolescents. Although African American teens make up only 15% of the adolescent population in the U.S., they account for about two thirds of new AIDS cases among teens. An Atlanta, Georgia study involving a population composed primarily of urban African American teens demonstrated that few of the teens who tested positive for HIV were aware of the risks involved in sexual activity. Because of this population's increased risk for contracting HIV and other STDs, prevention programs that specifically target African American teens are necessary. This study will evaluate the joint and separate effectiveness of two HIV/STD prevention programs, small group training and mass media messages, in providing protection against acquiring STDs and maintaining safer sex behavior.

African American adolescents will be recruited for this single-blind, 18-month study through community-based organizations in four different cities. All participants will first complete a computer-administered survey to assess sexual attitudes, beliefs, and behaviors. They will also provide a urine sample for STD testing. Following these baseline assessments, participants will be randomly assigned to either the Focus on Youth (FOY) HIV prevention program or the Promoting Health Among Teens general health intervention. Both programs will involve eight 1-hour small group sessions that will occur over three Saturdays. Participants in the FOY program will learn safe sex and abstinence skills. Participants in the Promoting Health Among Teens intervention will receive general health information about diet, substance use, and appropriate screening for common health conditions other than STDs. All participants who test positive for an STD during the study will receive treatment. Follow-up assessments will occur at Months 6, 12, and 18 post-intervention to determine program effectiveness.

The second prevention program, mass media messages, will be administered among all participating African American teens in one of the two participating Northern cities and one of the two participating Southern cities. Cities that will receive the media intervention will be randomly selected. The other city in each pair will serve as a control city. Tailored HIV/STD prevention messages will be delivered through local mass media. Telephone interviews will be conducted over a 34-month period among 900 randomly selected teens from both media and non-media cities to assess community-wide effectiveness of the program.

ELIGIBILITY:
Inclusion Criteria:

* Currently resides in one of the test cities

Exclusion Criteria:

* Presence of mental impairments

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1650 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
STD incidence | Measured at Months 6, 12, and 18 post-treatment

SECONDARY OUTCOMES:
Number of unprotected sexual occasions | Measured at Months 6, 12, and 18 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Romer, PhD, Principal Investigator — University of Pennsylvania; Ralph DiClemente, PhD, Principal Investigator — Emory University; Lawrence Brown, MD, Principal Investigator — Brown University; Peter Vanable, PhD, Principal Investigator — Syracuse University; Robert Valois, PhD, Principal Investigator — University of South Carolina
Locations (4):
- United States (4):
  - Emory University, Rollins School of Public Health, Atlanta, Georgia
  - Syracuse University, Department of Psychology, Syracuse, New York
  - Brown University, Rhode Island Hospital, Providence, Rhode Island
  - University of South Carolina, Arnold School of Public Health, Columbia, South Carolina

REFERENCES:
- [Derived] Foley JD, Vanable PA, Brown LK, Carey MP, DiClemente RJ, Romer D, Valois RF. Depressive symptoms as a longitudinal predictor of sexual risk behaviors among African-American adolescents. Health Psychol. 2019 Nov;38(11):1001-1009. doi: 10.1037/hea0000780. Epub 2019 Aug 5. PMID 31380687
- [Derived] Hennessy M, Romer D, Valois RF, Vanable P, Carey MP, Stanton B, Brown L, DiClemente R, Salazar LF. Safer sex media messages and adolescent sexual behavior: 3-year follow-up results from project iMPPACS. Am J Public Health. 2013 Jan;103(1):134-40. doi: 10.2105/AJPH.2012.300856. Epub 2012 Nov 15. PMID 23153149